CLINICAL TRIAL: NCT02068716
Title: Optimizing Prevention of Healthcare-Acquired Infections After Cardiac Surgery
Acronym: HAI
Status: Completed | Type: Observational
Sponsor: Dr. Donald Likosky (Other)
Collaborators: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Responsible Party: Sponsor-Investigator, Dr. Donald Likosky, Associate Professor, University of Michigan
Organization: University of Michigan (Other)
Other Study IDs: HAI_Umich; 2004-0428 (Other: UMichigan's IRB)
Record Dates: First submitted 2014-02-19; First posted 2014-02-21 (Estimated); Last update posted 2018-10-23 (Actual); Status verified 2018-10

CONDITIONS: Healthcare Associated Infectious Disease; Sternal Superficial Wound Infection; Sepsis; Pneumonia; Deep Sternal Infection
Keywords: Healthcare acquired infections; Cardiovascular Surgery; Mediastinitis; Thoracotomy; Conduit harvest or cannulation site
MeSH Terms: conditions — Cross Infection; Sepsis; Pneumonia; Mediastinitis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Adults with HAIs: Adult cardiac surgery patients who develop infections in hospitals within 30 days post surgery.
  We will exclude patients presenting with endocarditis.

SUMMARY:
Our Aim is to identify patient risk factors and clinical practices associated with healthcare-acquired infections (HAIs) after cardiac surgery.

We will use prospectively collected data housed within the MSTCVS-QC (Michigan Society of Thoracic & Cardiovascular Surgeons Quality Collaborative) to reveal risk factors that elevate a patient's risk of developing HAIs. The results of this analysis will form the foundation for the development of standardized regional practices to reduce HAIs. We will explore the effect of traditional patient-level measures (age, sex, comorbid conditions), process measures (timing and selection of antibiotics, continuous insulin infusion, transfusions), and surgical practices (use of bilateral internal mammary artery usage among diabetics, vein harvesting approach).

DETAILED DESCRIPTION:
More than 400,000 coronary artery bypass grafting (CABG) procedures are performed every year in the United States (U.S.). Patients undergoing CABG surgery are at risk for a number of adverse sequelae, many of which impact survival and contribute to overall health-care costs. Healthcare-acquired infections (HAIs), including pneumonia and superficial and deep sternal wound infections, occur among 16% of CABG patients and elevate a patient's risk of mortality and add excess upfront and long-term expenditures to the health care system.

A number of barriers prevent wide-scale improvements in HAl rates within the setting of CABG surgery. While a number of HAl prophylaxis measures have been developed, these measures do not fully encompass the set of practices that may impact a patient's risk of HAl. Identifying cardiac surgery specific risk factors would serve as the foundation for targeted quality improvement strategies. In the absence of definitive data concerning best practices, HAl prophylaxis is variable across surgeons and institutions, resulting in unnecessary morbidity and cost. Prior work has shown the value of implementing evidence-based protocols in the general intensive care unit setting. To what extent the implementation of cardiac surgery specific standardized practices results in lower HAl rates is uncertain. An understanding of the effectiveness of this approach would certainly assist surgeons and institutions in providing safer care to their patient populations.

Rates of HAIs vary from 0-26% across the 33 institutions performing CABG surgery in Michigan. This application seeks to reduce this rate by identifying and subsequently implementing standardized practices, and evaluating their impact on HAl rates. This study will be based on the prospective data and regional quality improvement activities and infrastructure of the Michigan Society of Thoracic and Cardiovascular Surgeons Quality Collaborative (MSTCVS-QC). We will evaluate the effectiveness of these standardized practices in reducing HAIs regionally and relative to national rates during the same time period.

Our Aim is to identify patient risk factors and clinical practices associated with HAIs after cardiac surgery.

We will use prospectively collected data housed within the MSTCVS-QC to reveal risk factors that elevate a patient's risk of developing HAIs. The results of this analysis will form the foundation for the development of standardized regional practices to reduce HAIs. We will explore the effect of traditional patient-level measures (age, sex, comorbid conditions), process measures (timing and selection of antibiotics, continuous insulin infusion, transfusions), and surgical practices (use of bilateral internal mammary artery usage among diabetics, vein harvesting approach).

ELIGIBILITY:
Inclusion Criteria:

* Female and male adult patients 18 and over undergoing cardiac surgery within the state of Michigan from January 1, 2011 through June 30, 2013.

Exclusion Criteria:

* Pregnant women,
* children,
* endocarditis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing adult cardiac surgery
Sampling Method: Non-Probability Sample
Enrollment: 911754 (Actual)
Dates: Start 2014-03; Primary Completion 2018-09-29 (Actual); Study Completion 2018-09-29 (Actual)

PRIMARY OUTCOMES:
Percent of patients having a healthcare-acquired infection (HAIs) post cardiac surgery. | In-hospital or within the first 30 days (for surgical infections) after surgery
  Overall HAIs include pneumonia, sepsis/septicemia, and surgical site infections, including deep sternal wound, thoracotomy, and harvest/cannulation site infections.

CONTACTS AND LOCATIONS:
Overall Officials: Donald S Likosky, Ph.D., Principal Investigator — University of Michigan
Locations (1):
- Mstcvs-Qc, Ann Arbor, Michigan, United States

REFERENCES:
- [Result] Shih T, Zhang M, Kommareddi M, Boeve TJ, Harrington SD, Holmes RJ, Roth G, Theurer PF, Prager RL, Likosky DS; Michigan Society of Thoracic and Cardiovascular Surgeons Quality Collaborative. Center-level variation in infection rates after coronary artery bypass grafting. Circ Cardiovasc Qual Outcomes. 2014 Jul;7(4):567-73. doi: 10.1161/CIRCOUTCOMES.113.000770. Epub 2014 Jul 1. PMID 24987052
- [Result] Likosky DS, Wallace AS, Prager RL, Jacobs JP, Zhang M, Harrington SD, Saha-Chaudhuri P, Theurer PF, Fishstrom A, Dokholyan RS, Shahian DM, Rankin JS; Michigan Society of Thoracic and Cardiovascular Surgeons Quality Collaborative. Sources of Variation in Hospital-Level Infection Rates After Coronary Artery Bypass Grafting: An Analysis of The Society of Thoracic Surgeons Adult Heart Surgery Database. Ann Thorac Surg. 2015 Nov;100(5):1570-5; discussion 1575-6. doi: 10.1016/j.athoracsur.2015.05.015. Epub 2015 Aug 28. PMID 26321440
- [Result] Strobel RJ, Liang Q, Zhang M, Wu X, Rogers MA, Theurer PF, Fishstrom AB, Harrington SD, DeLucia A 3rd, Paone G, Patel HJ, Prager RL, Likosky DS; Michigan Society of Thoracic and Cardiovascular Surgeons Quality Collaborative. A Preoperative Risk Model for Postoperative Pneumonia After Coronary Artery Bypass Grafting. Ann Thorac Surg. 2016 Oct;102(4):1213-9. doi: 10.1016/j.athoracsur.2016.03.074. Epub 2016 Jun 1. PMID 27261082
- [Result] Brescia AA, Rankin JS, Cyr DD, Jacobs JP, Prager RL, Zhang M, Matsouaka RA, Harrington SD, Dokholyan RS, Bolling SF, Fishstrom A, Pasquali SK, Shahian DM, Likosky DS; Michigan Society of Thoracic and Cardiovascular Surgeons Quality Collaborative. Determinants of Variation in Pneumonia Rates After Coronary Artery Bypass Grafting. Ann Thorac Surg. 2018 Feb;105(2):513-520. doi: 10.1016/j.athoracsur.2017.08.012. Epub 2017 Nov 23. PMID 29174785
- [Derived] Likosky DS, Harrington SD, Cabrera L, DeLucia A 3rd, Chenoweth CE, Krein SL, Thibault D, Zhang M, Matsouaka RA, Strobel RJ, Prager RL. Collaborative Quality Improvement Reduces Postoperative Pneumonia After Isolated Coronary Artery Bypass Grafting Surgery. Circ Cardiovasc Qual Outcomes. 2018 Nov;11(11):e004756. doi: 10.1161/CIRCOUTCOMES.118.004756. PMID 30571334